CLINICAL TRIAL: NCT01928225
Title: A Randomized, Placebo-controlled Trial of Pre-treatment HPV Vaccination on Outcomes to LEEP Treatment of Cervical High Grade Squamous Intraepithelial Lesions in HIV-infected Women.
Brief Title: Randomized, Double Blind Trial of the Quadrivalent HPV Vaccine to Improve Responses to LEEP Treatment of Cervical HSIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Cynthia S Firnhaber, Technical Director of the Clinical HIV Research Unit, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QHPV-RTC
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Cervical High Grade Squamous Intraepithelial Lesion
Keywords: HSIL; CIN; HPV; HPV vaccination; gardasil; HIV; cervical dysplasia; LEEP; cervical cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Papillomavirus vaccine (Experimental): Participants receive the experimental quadrivalent Human Papillomavirus vaccine at entry, week 4 and week 26.
  Interventions: Biological: Human Papillomavirus vaccine
- Saline placebo (Placebo Comparator): The participants receive saline placebo at entry, week 4 and week 26.
  Interventions: Biological: Human Papillomavirus vaccine

INTERVENTIONS:
Biological: Human Papillomavirus vaccine — The participants receive the qHPV vaccine at entry, week 4 and week 26
  Other Names: qHPV vaccine

SUMMARY:
Cervical cancer occurs commonly in HIV-infected women in South Africa. These women have poor response to treatment of cervical cancer precursors. This study will test whether giving the quadrivalent vaccine to women prior to surgical treatment of the cervical cancer precursor will improve outcomes. We hypothesize that pre-treatment HPV vaccine will result in a reduced occurrence or cervical cancer precursors in follow-up.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blinded, placebo-controlled, phase II trial of the quadrivalent human papillomavirus vaccine (qHPV) in HIV-infected women to prevent occurrence of cervical HSIL after LEEP/LLETZ. Participants will undergo colposcopy with directed biopsies, cervical cytology, and stored HPV testing prior to vaccination. Participants will be randomized to the quadrivalent vaccine or saline placebo to be given at entry, week 4, and week 26. Women will have LEEP treatment at week 4. Participants will be seen in follow-up for cervical cytology, colposcopy with directed biopsies at weeks 26 and 52, and stored HPV specimens. Treatment assignment will be unblinded after study follow-up is completed for the last study participant. Women aged 45 or less randomized to placebo will be offered open label HPV vaccine after the study is concluded..

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection
2. Women aged ≥ 18 years.
3. Cervical HSIL on biopsy (i.e. CIN2 and/or CIN3)
4. For participants of reproductive potential, negative serum or urine pregnancy test
5. All study participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or in vitro fertilization) during study participation (from the time of study entry until week 52).

Exclusion Criteria:

1. History or current biopsy diagnosis of invasive or microinvasive cervical, vaginal, vulvar, anal or oropharyngeal cancer
2. Prior hysterectomy
3. Cervical cryotherapy or LEEP/LEETZ within one year of entry.
4. Cervical, vulvar, or vaginal lesions suspicious for cancer, unless biopsies show no invasive cancer
5. Prior receipt of one or more doses of an HPV vaccine.
6. Receipt of anticoagulants other than aspirin or nonsteroidal anti-inflammatory drugs (NSAIDS) within 14 days prior to entry.
7. Known allergy/sensitivity or any hypersensitivity to yeast or any of the components of the study product or its formulation (see section 5.2 for a list of components).
8. Hemophilia or other bleeding diatheses.
9. Use of any systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids, other than inhaled corticosteroids or prednisone ≤ 10 mg (or equivalent) , investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry.
10. Breastfeeding
11. Less than 3 months post-partum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Wilkin, M.D. MPH, Study Chair — Weill Medical College of Cornell University; Cynthia Firnhaber, M.D., Study Chair — University or Witswatersrand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Firnhaber C, Swarts A, Jezile V, Mulongo M, Goeieman B, Williams S, Faesen M, Michelow P, Wilkin T. Human Papillomavirus Vaccination Prior to Loop Electroexcision Procedure Does Not Prevent Recurrent Cervical High-grade Squamous Intraepithelial Lesions in Women Living With Human Immunodeficiency Virus: A Randomized, Double-blind, Placebo-controlled Trial. Clin Infect Dis. 2021 Oct 5;73(7):e2211-e2216. doi: 10.1093/cid/ciaa1456. PMID 32975556

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Human Papillomavirus Vaccine | Saline Placebo
Started | 90 | 90
Completed | 87 | 87
Not Completed | 3 | 3
Not completed — Pregnancy | 1 | 0
Not completed — basaloid cervical cancer | 1 | 0
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Human Papillomavirus Vaccine: Participants receive the quadrivalent Human Papillomavirus vaccine at entry, week 4 and week 26.
- Total: Total of all reporting groups
Arm/Group | Human Papillomavirus Vaccine | Saline Placebo | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40.1 [34.8 to 46.6] | 39.1 [35.2 to 44.2] | 39.2 [34.9 to 45.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 90 | 180
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 90 | 90 | 180
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 90 | 86 | 176
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  South Africa | 90 | 90 | 180
HSIL/ASC-H cervical cytology [Count of Participants; unit: Participants] — HSIL= high grade squamous intraepithelial lesions; ASC-H=atypical squamous cells suggestive of HSIL
  Participants | 86 | 83 | 169
Plasma HIV-1 RNA <200 copies/mL [Count of Participants; unit: Participants] — Population: Plasma HIV RNA was missing on 17 participants
  Participants
    number analyzed (Participants) | 81 | 82 | 163
    (all) | 77 | 76 | 153
CD4 [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: CD4 cell counts were missing on 17 participants
  cells/mm^3
    number analyzed (Participants) | 81 | 82 | 163
    (all) | 511 [300 to 689] | 483 [337 to 745] | 489 [302 to 724]
Nadir CD4 [Median (Inter-Quartile Range); unit: cells/mm3] — Population: Nadir CD4 counts were not available for two participants
  cells/mm3
    number analyzed (Participants) | 89 | 89 | 178
    (all) | 125 [61 to 200] | 108 [50 to 200] | 116 [50 to 200]

OUTCOME MEASURES:

1. Primary Outcome: Cervical HSIL
Description: For this trial, the primary endpoint is high-grade squamous intraepithelial lesions (HSIL) or atypical squamous cells suggestive of HSIL found on cervical cytology, or HSIL found on cervical biopsy specimens at either the week 26 or week 52 visit.
Time Frame: up to 52 weeks
Population: Six participants did not have cytologic or histologic samples available for the primary endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Human Papillomavirus Vaccine | Saline Placebo
Number analyzed (Participants) | 87 | 87
Participants | 46 | 39
Statistical Analysis 1: Comparison: Human Papillomavirus Vaccine vs Saline Placebo; Test type: Superiority; p = .29, Chi-squared — <0.05 was considered statistically significant; Risk Ratio (RR) = 1.18, 95% CI 2-sided [.87 to 1.6]

2. Secondary Outcome: Cervical Cytology
Description: Cervical cytology abnormalities according to the Bethesda scale. The Bethesda scale classifies cytologic abnormalities. We have dichotomized the outcomes into high grade squamous intraepithelial lesions (HSIL)/atypical squamous cells suggestive of HSIL, or no evidence of intraepithelial lesions or malignancy (NILM)/atypical squamous cells of unknown significance (ASC-US)/low grade squamous intraepithelial lesions (LSIL). We report the number of women in each category.
Time Frame: Week 26
Population: Comparison of cytologic outcomes between arms at week 26. Nine participants are missing due to a missed visit, loss to follow-up, or unsatisfactory cytology result.
Measure: Count of Participants; unit: Participants
Groups:
- Human Papillomavirus Vaccine: Participants receive the experimental Human Papillomavirus vaccine at entry, week 4 and week 26.
Arm/Group | Human Papillomavirus Vaccine | Saline Placebo
Number analyzed (Participants) | 86 | 85
Participants
  HSIL or ASC-H | 34 | 26
  NILM/ASCUS/LSIL | 52 | 59
Statistical Analysis 1: Comparison: Human Papillomavirus Vaccine vs Saline Placebo; Test type: Superiority; p = .22, Chi-squared; Risk Ratio (RR) = 1.26, 95% CI 2-sided [.85 to 1.95]

ADVERSE EVENTS:
Time Frame: one year
Description: Grade 3 or 4 adverse event related to study vaccination. Please note that only deaths, serious adverse events, and grade 3 or 4 adverse events related to study vaccination were captured. Other grade 3 or 4 events were not captured per protocol. Grade 1 or 2 adverse events were not captured per protocol.
Arm/Group | Human Papillomavirus Vaccine | Saline Placebo
All-Cause Mortality (participants affected / at risk) | 1/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 2/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Papillomavirus Vaccine (N=90) | Saline Placebo (N=90)
death (Cardiac disorders) | 1 (1) | NA — Death of unknown cause
cervical cancer (Reproductive system and breast disorders) | 1 (90) | NA — Basaloid Cervical Cancer

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT01928225/Prot_SAP_000.pdf